CLINICAL TRIAL: NCT02634437
Title: A Single-Dose, Open-Label, Pharmacokinetic Study Of Ulipristal Acetate In Healthy Subjects With Normal Renal Function And Patients With Moderately Or Severly Impaired Renal Function
Brief Title: Study of Ulipristal Acetate in Female Patients With Moderately or Severely Impaired Renal Function, Compared With Matched Healthy Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UPA-PK-02
Record Dates: First submitted 2015-12-16; First posted 2015-12-18 (Estimated); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Renal Function
MeSH Terms: interventions — ulipristal acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Normal Renal Function (Experimental): Ulipristal acetate, 10 mg, oral administration
  Interventions: Drug: Ulipristal acetate
- Moderate Renal Impairment (Experimental): Ulipristal acetate, 10 mg, oral administration
  Interventions: Drug: Ulipristal acetate
- Severe Renal Impairment (Experimental): Ulipristal acetate, 10 mg, oral administration
  Interventions: Drug: Ulipristal acetate

INTERVENTIONS:
Drug: Ulipristal acetate

SUMMARY:
This study is designed to observe the effect of renal function on the pharmacokinetic, safety, and tolerability profiles of Ulipristal acetate following administration of a single oral dose of a 10 mg Ulipristal acetate tablet.

ELIGIBILITY:
Inclusion Criteria for Patients with Renal Impairment:

* Have a negative result from a serum pregnancy test at screening and a negative result from a serum or urine pregnancy test on Day -1
* If premenopausal, have regular menstrual cycles (cycles of 24-35 days duration) over the past 6 months as reported by the patient
* If female of childbearing potential, agree to use an effective method of contraception (i.e., condom plus diaphragm with spermicide, condom with spermicide, or nonhormonal intrauterine device) and not become pregnant throughout the study. Subjects who are at least 2-years postmenopausal (with supporting documentation from an obstetrician/gynecologist) or who have had tubal ligation or hysterectomy will not be considered to be of childbearing potential
* Be nonsmoking (never smoked or have not smoked within the previous 6 months) or a light smoker (fewer than 10 cigarettes per day within the previous 3 months)
* For Patients with Renal Impairment, have medical history, physical examination, laboratory, and other test results consistent with their degree of renal impairment, as determined by the Investigator
* For Patients with Normal Renal Function, have a state of general good health based on medical history and routine physical examination and are matched to the age and weight of the renal dysfunction patients (mean group difference ±10 years for age and < 20% for weight)

Exclusion Criteria:

* Known hypersensitivity to Ulipristal Acetate (UPA) or other selective progesterone receptor modulators
* For Patients with Renal Impairment, clinically significant disease state, in the opinion of the examining physician, in any body system (other than renal function impairment)
* For Patients with Normal Renal Function, clinically significant disease state, in the opinion of the examining physician, in any body system
* Positive test results for anti-human immunodeficiency virus type 1, hepatitis B surface antigen, or anti-hepatitis C virus at screening
* Abnormal and clinically significant results on physical examination, medical history, serum chemistry, hematology, or urinalysis
* History of alcohol or other substance abuse within the previous 5 years
* Positive test results for benzoylecgonine (cocaine), methadone, barbiturates, amphetamines, benzodiazepines, alcohol, cannabinoids, opiates, or phencyclidine at screening or Day -1. Patients with Renal Impairment many be enrolled if the positive test result is due to prescription drug use and approved by the Principal Investigator and Sponsor Study Physician, on a case-by-case basis
* Participation in any other clinical investigation using an experimental drug requiring repeated blood or plasma draws within 30 days of IP administration
* Participation in a blood or plasma donation program within 60 or 30 days, respectively, of Investigational Product (IP) administration
* Previously participated in an investigational study of Ulipristal Acetate
* Breastfeeding

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2016-12-09 (Actual); Study Completion 2016-12-09 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve of ulipristal acetate from time 0 to time t (AUC 0-t) | Day 1 (0 hour) to Day 8 (168 hours)
Maximum plasma drug concentration (Cmax) of ulipristal acetate | Day 1 (0 hour) to Day 8 (168 hours)
Time of maximum plasma drug concentration (Tmax) of ulipristal acetate | Day 1 (0 hour) to Day 8 (168 hours)
Terminal elimination half-life (T½) of ulipristal acetate | Day 1 (0 hour) to Day 8 (168 hours)
Apparent total body clearance of ulipristal acetate from plasma after extravascular administration (CL/F) of ulipristal acetate | Day 1 (0 hour) to Day 8 (168 hours)
Apparent volume of distribution during the terminal phase after extravascular administration (Vz/F) of ulipristal acetate | Day 1 (0 hour) to Day 8 (168 hours)
Area under the plasma concentration versus time curve of ulipristal acetate from time 0 to infinity (AUC 0-∞) | Day 1 (0 hour) to Day 8 (168 hours)

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve of PGL4002 (ulipristal acetate active metabolite) from time 0 to time t (AUC 0-t) | Day 1 (0 hour) to Day 8 (168 hours)
Time of maximum plasma drug concentration (Tmax) of PGL4002 (ulipristal acetate active metabolite) | Day 1 (0 hour) to Day 8 (168 hours)
Terminal elimination half-life (T½) of PGL4002 (ulipristal acetate active metabolite) | Day 1 (0 hour) to Day 8 (168 hours)
Maximum plasma drug concentration (Cmax) of PGL4002 (ulipristal acetate active metabolite) | Day 1 (0 hour) to Day 8 (168 hours)
Cumulative amount of ulipristal acetate excreted into urine from time zero to time t (Ae0-t) | Day 1 (0 hour) to Day 8 (168 hours)
Renal clearance of ulipristal acetate from plasma (CLR) | Day 1 (0 hour) to Day 8 (168 hours)
Percent of dose excreted as unchanged ulipristal acetate in urine (%Dose) | Day 1 (0 hour) to Day 8 (168 hours)
Cumulative amount of PGL4002 excreted into urine from time zero to time t (Ae0-t) | Day 1 (0 hour) to Day 8 (168 hours)
Renal clearance of PGL4002 from plasma (CLR) | Day 1 (0 hour) to Day 8 (168 hours)
Area under the plasma concentration versus time curve of PGL4002 (ulipristal acetate active metabolite) from time 0 to infinity (AUC 0-∞) | Day 1 (0 hour) to Day 8 (168 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Laishun Chen, Study Director — Forest Laboratories Inc, an affiliate of Allergan plc
Locations (5):
- United States (5):
  - Division of Clinical Pharmacology, University of Miami, Miami, Florida
  - Clinical Pharmacology of Miami, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Prism Clinical Research, Saint Paul, Minnesota
  - QPS Bio-Kinetic, Springfield, Missouri